CLINICAL TRIAL: NCT06723015
Title: Study of Tau PET Outcomes in Patients Receiving Anti-amyloid Immunotherapies
Brief Title: Tau PET Outcomes With Anti-amyloid Immunotherapies
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Petrice M. Cogswell, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24-004371
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Impairment, Mild; Dementia, Mild; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Lymphoma, Follicular; Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Untreated historical controls enrolled in Mayo Clinic Study of Aging (IRB 14-004401), Mayo Alzheimer's Disease Research Center (IRB 712-98), and Brain Amyloid Imaging with Pittsburgh Compound B in Normal Aging, Mild Cognitive Impairment, and Dementia (IRB 08-005553).
- Treatment Group (Experimental): Subjects with a diagnosis of mild cognitive impairment (MCI) or mild dementia due to Alzheimer's disease and amyloid positive, who are starting anti-amyloid immunotherapy.
  Interventions: Drug: 18F-AV-1451

INTERVENTIONS:
Drug: 18F-AV-1451 — Subjects will receive two Tau PET (18F--AV-1451) brain scans with approximately 10 mCi (370 MBq) (+/- 10%mCi) of 18F-AV-1451. Images will be collected for a 20-minute acquisition between 80-100 minutes after injection.
  Tau PET scans will occur at baseline and 12-18 months after completing anti-amyloid immunotherapy treatment..
  Arms: Treatment Group

SUMMARY:
This is an imaging study of patients with mild Alzheimer's disease receiving amyloid-targeting therapy and under the care of neurologists at Mayo Clinic in Rochester, MN.

ELIGIBILITY:
Inclusion Criteria

* Age 50-90 years
* Male or female
* Mild cognitive impairment due to AD or mild AD
* Amyloid positive via CSF or PET
* Meets other eligibility criteria for anti-amyloid immunotherapy
* Subject or delegate provides informed consent

Exclusion Criteria

* Subjects unable to lie down without moving for 10 minutes.
* Women who are pregnant or cannot stop breast feeding for 24 hours.
* Claustrophobic patients unable to tolerate the scans (no sedation can be offered).

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change in tau PET Standardized Uptake Value (SUVR) | Baseline, 18 months
  A PET Standardized Uptake Value (SUV) is measured by calculating the ratio of the radioactivity concentration within a specific region of interest (ROI) on a PET scan, divided by the injected dose of the radiotracer per unit of the patient's body weight. The calculated Standardized Uptake Value (SUVR) is reported as a single number, with higher values indicating greater tracer uptake in the target region relative to the reference region

SECONDARY OUTCOMES:
Number of subjects to develop amyloid-related imaging abnormalities (ARIA) | 18 months
  ARIA is defined as edema (parenchymal edema or sulcal effusion, ARIA-E) and hemorrhage (microhemorrhages and superficial siderosis, ARIA-H). ARIA is detected on the patient's routine clinical brain MRIs.

CONTACTS AND LOCATIONS:
Overall Officials: Petrice Cogswell, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No